CLINICAL TRIAL: NCT01584635
Title: Peroral Endoscopic Myotomy (POEM) for Treatment of Achalasia
Brief Title: The Role That Peroral Endoscopic Myotomy (POEM) Could Play in the Treatment of Achalasia
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David A. Katzka, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-005252
Record Dates: First submitted 2012-01-12; First posted 2012-04-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Achalasia
Keywords: Less invasive treatment for Achalasia
MeSH Terms: conditions — Esophageal Achalasia | interventions — Heller Myotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peroral Endoscopic Myotomy (POEM) (Experimental): Peroral Endoscopic Myotomy- a less invasive treatment for patients with Achalasia
  Interventions: Procedure: Peroral Endoscopic Myotomy a less invasive treatment for Achalasia

INTERVENTIONS:
Procedure: Peroral Endoscopic Myotomy a less invasive treatment for Achalasia — In this study we will follow patients undergoing Peroral Endoscopic Myotomy at 1 and 6 months post surgery,1,2,3,4,and 5 years post surgery with esophageal high resolution Manometry and a Barium Esophagram when it is not standard of care. We will have you fill out a symptom questionnaire at each visit
  Other Names: Achalasia; Heller myotomy; Dysphagia; Peroral Endoscopic Myotomy; Disease of the muscle of the esophagus.; Disorder of the swallowing tube.; Esophageal Motility Disorders; Esophageal Achalasia

SUMMARY:
Based on the work of the Doctors at the Mayo Clinic Rochester, a new technique for a less invasive treatment for Achalasia has been developed.

The purpose of this study is to decide the role this less invasive treatment (Peroral Endoscopic Myotomy) has in the treatment of patient's with achalasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 80 with achalasia diagnosed by a combination of compatible symptoms, barium esophagography and high resolution manometry.

Exclusion Criteria:

* Patients who are poor surgical risks, have had previous treatment for achalasia or esophageal or gastric surgery, have an epiphrenic diverticulum or are unwilling to be followed in the protocol.
* Female patients are eligible if they are NOT pregnant or lactating AND ne of the following criteria is met:
* The patient is surgically sterile (by means of hysterectomy/bilateral tubal ligation)
* The patient is at least one year postmenopausal (no menses for 12 months).
* The patient is using a highly effective method of contraception, if childbearing potential, AND has a negative urine human chorionic gonadotropin beta subunit (ß HCG) pregnancy test result during Screening, and prior to trial drug administration.
* Highly effective methods of birth control are defined as those which result in a low failure rate when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomized partner.
* Withdrawal, single- or double barrier methods (including condoms) and rhythm methods are NOT ACCEPTABLE methods of contraception for the purposes of this clinical trial due to the high incidence of contraceptive failures with these methods.
* Vulnerable populations, such as those with diminished mental acuity, will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 5 years post surgery
  Patients in this study, undergoing the Peroral Endoscopic Myotomy treatment for Achalasia, will be accessed at 1 month, 6 months, at 1-2-3-4 and year 5 post surgery. We will measure outcomes by number of adverse events, Eckardt symptom score, barium esophagram, and manometry studies.

SECONDARY OUTCOMES:
Eckardt symptom score | 5 years
  By following participants regularly and closely both by symptomatic and objective criteria, we will be able to determine factors that predict response to the POEMS procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David Katzka, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States